CLINICAL TRIAL: NCT05225870
Title: Enhanced Cortactin Expression is Associated With Increased Tumor Invasiveness and Nodal Metastasis in Egyptian Patients With Colorectal Adenocarcinomas
Brief Title: Significance of Cortactin Expression in Colorectal Adenocarcinomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Maisa Hashem Mohammed, Lecturer of Pathology, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Soh-Med-22-01-33
Record Dates: First submitted 2022-01-23; First posted 2022-02-07 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Cancer Colon
Keywords: cancer colon; Cortactin; Immnuohistochemistry
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Fifty, paired formalin-fixed and paraffin embedded tissue blocks from the colorectal carcinomas and adjacent non neoplastic colonic mucosa will be prepared and sectioned. From each block; one section will be stained by Haematoxaline and Eosine to establish diagnosis of colorectal carcinomas and to determine the degree of differentiation and degree of invasion of the underlying colonic tissues. Corresponding sections from each Formalin-fixed paraffin embedded tissue blocks will be immunohistochemically stained by anti- Human Cortactin antibody, to detect any association between cortactin expression and colorectal carcinoma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with colorectal carcinoma (Other): patients with colorectal carcinoma will undergo colectomy. their colectomy specimens will be sectioned, tissue blocks will be prepared from tumor and adjacent normal mucosa. sections will be stained immunohistochemically by antibody against cortactin.
  Interventions: Genetic: immunohistochemical staining

INTERVENTIONS:
Genetic: immunohistochemical staining — sections from colorectal carcinoma will be immunohistochemically stained by anti-Cortactin antobody.

SUMMARY:
Colorectal carcinoma is one of the most aggressive malignant epithelial neoplasms affecting the gastrointestinal tract. The incidence of colorectal carcinoma is obviously increasing in developing countries, where the physical inactivity and the consumption of animal fat-rich food became more evident. Colorectal tumorigenesis is a multistep process which is initiated by adenoma and is terminated by carcinoma, the latter shows variable degrees of tumor differentiation and invasiveness. During the adenoma-carcinoma process; a series of genetic mutations occur. Detection of these genetic mutations will help in the development of novel therapeutic agents, which in turn will improve patients' outcomes. Cortactin (CTTN) is a Src kinase substrate, encoded by a gene located on chromosome 11. CTTN binds to and activates Arp 2/3 and stabilizes the dynamic actin assembly after its formation. So, it become clear that CTTN is involved in the formation of the leading-edges cellular protrusions.

DETAILED DESCRIPTION:
Colorectal carcinoma is a highly lethal malignant epithelial tumor involving humans. The incidence of colorectal carcinoma is steadily increasing in developing countries, this could be assigned to low physical activity together with high consumption of animal fat-rich food. malignancy of the colon is a multistep process which is initiated by adenoma that proceeds to carcinoma, the latter includes a wide variety of tumor phenotypes. During the adenoma-carcinoma process; a series of genetic and epigenetic alterations occur. Detection of these genetic alterations is of great benefit in the future management of colorectal carcinomas. Cortactin (CTTN) is a Src kinase substrate, encoded by a gene located on chromosome 11. CTTN anchors the dynamic actin assembly . CTTN is implicated in the formation of the leading-edges cellular protrusions.the aim of this study is to evaluate expression of CTTN in 50 cases of colorectal adenocarcinomas and their adjacent normal colonic mucosae.

ELIGIBILITY:
Inclusion Criteria:

* patients with colorectal carcinomas who underwent colectomy operations.

Exclusion Criteria:

* specimens obtained by lower endoscopy only, patients who received pre-operative chemotherapy.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
immunohistochemical evaluation of Cortactin expression | 8 weeks
  Fifty patients with colorectal adenocarcinoma will be enrolled in the study. Formalin-fixed and paraffin embedded tissue blocks will be prepared from the tumor and adjacent normal colorectal mucosa in the Pathology lab. Sections will be stained by Hematoxalin and Eosin to diagnose the tumor phenotype. Additional sections will be mounted on coated slides and stained immunohistochemically by antibodies against human Cortactin . immunohistochemical expression of Cortactin will be evaluated in both the tumor sections and adjacent normal mucosa by using Immuno-reactive score. Expression of Cortactin in tumor tissues will be statistically correlated to degree of tumor differentiation, tumor invasion and nodal metastasis.

CONTACTS AND LOCATIONS:
Overall Officials: Maisa H Mohammed, Principal Investigator — a lecturer of pathology, Sohag faculty of medicine
Locations (1):
- Maisa Hashem Mohammed, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No